CLINICAL TRIAL: NCT03539094
Title: Randomized Controlled Trial on Intermittent Fasting in Multiple Sclerosis
Brief Title: Intermittent Fasting in Multiple Sclerosis
Acronym: IFMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201707010
Record Dates: First submitted 2018-04-27; First posted 2018-05-29 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Intermittent fasting; western diet; microbiome
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the intervention because they will not know the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (Experimental): The subjects randomized to this group will do IF by restricting their diet and consuming few calories two days per week. During the days of fasting, subjects will be allowed to drink water, calorie-free beverages, and eat fresh, steamed or roasted non-starchy vegetables.
  Interventions: Other: Intermittent fasting
- Western diet (No Intervention): The subjects randomized to this group will eat a standard western style diet.

INTERVENTIONS:
Other: Intermittent fasting — the subjects randomized to this group will do IF by restricting their diet and consuming few calories two days per week. During the days of fasting, subjects will be allowed to drink water, calorie-free beverages, and eat fresh, steamed or roasted non-starchy vegetables.
  Arms: Intermittent fasting

SUMMARY:
This is a randomized controlled trial that will test the effects of intermittent fasting (IF) in subjects with relapsing-remitting MS (RRMS). The goal of this clinical trial is to acquire objective evidence regarding whether an IF diet has beneficial effects in MS patients.Two dietary regimens, IF and western diet, will be compared in a randomized, controlled, single-blinded 12 week trial in RRMS patients. This is a single-center study.

DETAILED DESCRIPTION:
RRMS patients will be enrolled in a randomized, controlled, single-blinded 12 week trial in which IF will be compared to a standard western diet. Patients will be recruited at the John L. Trotter MS center and randomly assigned to either a standard western diet or an IF diet (1:1). Enrolled subjects will complete a clinical and laboratory assessment before starting the diet (baseline), at week 6 and at end of the study (week 12). The primary outcome will be leptin at week 12 measured in the peripheral blood. Secondary outcomes will be: 1) peripheral blood metabolic profiling; 2) anthropometric (body mass index and waist circumference) and total body fat measures; 3) gut microbiota richness and composition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS (2010 Mc Donald criteria).
* EDSS <6.0 and disease duration ≤ 15 years.
* On an injectable therapy for MS, glatiramer acetate (GA) or beta-interferon (beta-IFN) for at least 3 months prior to the study and with no anticipated changes of the medication for the 12 week study duration.
* Age ≥18 years.
* BMI > 22 and < 35 kg/m2 with stable weight in the 3 months prior to screening.

Exclusion Criteria:

* History of any chronic disease process (excluding MS) that could interfere with interpretation of results.
* Diagnosis in the past of an eating disorder (anorexia, bulimia, or binge eating).
* Relapsing at the time of enrollment.
* On corticosteroid treatment (oral or intravenous) in the past month. Nasal corticosteroid treatments are allowed.
* Diagnosis of diabetes or at time of OGTT (fasting glucose >126 mg/dl or > 200 mg/dl at 2 hours with a load of 75 g of glucose
* History of food allergies or food intolerance that would interfere with the study.
* History of antibiotic treatment within the past 3 months prior to enrollment
* Use of anticoagulant drugs (like Warfarin or Coumadin) that need to monitor their intake of vegetables containing high levels of vitamin K.
* Currently on a special diet and not willing to stop at least one month prior to enrollment
* Currently taking omega 3/fish oil supplements and not willing to stop administration one month prior to enrollment
* Currently pregnant or plan to become pregnant within 6 months
* Current tobacco or e-cigarette smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Leptin | 12 weeks
  Leptin at week 12 measured in the peripheral blood

SECONDARY OUTCOMES:
Peripheral metabolic and inflammatory profiling | 12 weeks
  Adipokine and inflammatory markers at week 12 measured in the peripheral blood
Anthropometric measure | 12 weeks
  Weight and height will be combined to report BMI in kg/mg^2
Anthropometric measure | 12 weeks
  Waist circumference in centimeters
Gut microbiota | 12 weeks
  Gut microbiota richness and composition

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Ghezzi L, Tosti V, Shi L, Cantoni C, Mikesell R, Lancia S, Zhou Y, Obert K, Dula C, Sen MK, Ge A, Tolentino M, Bollman B, Don AS, Matarese G, Colamatteo A, La Rocca C, Lepore MT, Raji CA, Rahmani F, Wu GF, Naismith RT, Fontana L, Cross AH, Salter A, Piccio L. Randomised controlled trial of intermittent calorie restriction in people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2025 Jan 16;96(2):158-169. doi: 10.1136/jnnp-2024-333465. PMID 39137977